CLINICAL TRIAL: NCT02837822
Title: Effects of Spinal Cord Stimulation on Sensory Perceptions of Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Michel Prud'Homme, MD, PhD, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2015-2072
Record Dates: First submitted 2016-06-03; First posted 2016-07-20 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pain; Complex Regional Pain Syndrome; Failed Back Surgery Syndrome
Keywords: Spinal Cord Stimulation; Quantitative Sensory Testing
MeSH Terms: conditions — Chronic Pain; Complex Regional Pain Syndromes; Failed Back Surgery Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stimulation Off (Active Comparator): Patients receiving the intervention "implantation with a spinal cord stimulator". The system is turn Off during the experiment.
  Interventions: Device: Spinal cord stimulator; Procedure: Implantation of a spinal cord stimulator
- Stimulation On (Active Comparator): Patients receiving the intervention "implantation with a spinal cord stimulator". The system is turn On during the experiment.
  Interventions: Device: Spinal cord stimulator; Procedure: Implantation of a spinal cord stimulator

INTERVENTIONS:
Device: Spinal cord stimulator — Spinal cord stimulator is a reversible and minimally invasive neuromodulation device used for the treatment of various diseases related to chronic pain, including CRPS and FBSS. Briefly, this technology uses electrical pulses to generate action potentials in nerve cells that induce paresthesias (buzzing or tingling sensations) in the affected limb and can relieve pain.
  Other Names: Dorsal column stimulation
Procedure: Implantation of a spinal cord stimulator — The electrical pulses are induced by one or more electrodes surgically implanted into the epidural space. These electrodes are usually placed under the skin in the abdomen or upper buttock.

SUMMARY:
It's well known that Spinal cord stimulation (SCS) changes the perception of chronic pain in the area stimulated by epidural electrodes. However, we don't know the effect of this type of stimulation on the perception of external sensations (temperature, touch, pressure, and vibration) and sharp pain. Quantitative sensory testing (QST) is used to quantify somatosensory phenotype. This QST battery tests different subtypes of nerve fibres (Aβ, Aδ and C) involved in the transduction of sensory information from the periphery to the spinal cord.

The purpose of this study is to evaluate the effects of the SCS on sensory perceptions of patients with chronic pain (CRPS, FBSS). Sensorial perception tests will be carried out in accordance with a standardized procedure (Rolke et al. Pain, 2006). For non-implanted patients, an initial visit will be conducted before the operation. For all participants, two other visits will take place at least 6 months after the operation to perform the tests with and without stimulation.

DETAILED DESCRIPTION:
Spinal cord stimulation (SCS) is a reversible and minimally invasive neuromodulation technique employs for the treatment of chronic neuropathic pain. Even if SCS is an established technology for the management of complex regional pain syndrome (CRPS) and failed back surgery syndrome (FBSS), its impacts on the sensory perception system remain misunderstood.

The purpose of this study is to evaluate the effects of the SCS on sensory perceptions of patients with chronic pain (CRPS, FBSS). Sensorial perception tests will be carried out in accordance with a standardized procedure (Rolke et al. Pain, 2006) at the level of maximum pain area (painful leg), and at two non-painful areas (contralateral leg and ipsilateral arm). The thermode "Thermal Sensory Analyser TSA-II NeuroSensory Analyzer" and its complement "Vibratory Sensory Analyzer VSA-3000" (Medoc) will be used to assess warm, cold and vibratory detection thresholds, as well as heat and cold painful thresholds. Von Frey monofilaments (Bioseb) will be used to evaluate the mechanical detection threshold. The algometer "Force Ten ™ FDX Digital" (Wagner) will measure the pressure pain threshold. Dynamic mechanical allodynia will be assessed with a standardized brush (SENSELab Brush-05, Somedic). The Neuropen (Owen Mumford) will be used to test the temporal pain summation. Participants will be recruited through the neuromodulation clinic located in Enfant-Jésus Hospital (Québec, Canada).

For non-implanted patients, an initial visit will be conducted before the operation. For all participants, two other visits will take place at least 6 months after the operation to perform the tests with and without stimulation (the order of these visits will be randomized).

For each test, an average of the absolute differences (with-without stimulation) and its confidence interval will be calculated. The results will be considered significant with p values inferior to 0,05. All analyzes will be performed with SAS (SAS 9.3 Institute Inc, Cary, NC, USA).

The protocol was peer reviewed and approved by the Ethics Committee of Enfant-Jésus Hospital. All subjects will participate after written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a diagnosis of CRPS or FBSS that meet International Association for the Study of Pain's criteria;
* Pain in one leg;
* Paresthesia area limited to the treated leg;
* No changes in the programming patterns of the device for a minimum of 30 days before the tests;
* Informed consent.

Exclusion Criteria:

- Wounds or infections at the painful site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in sensory thresholds | Baseline and at least 6 months post-implantation
  Sensorial perception tests will be carried out in accordance with a standardized procedure (Rolke et al. Pain, 2006). The thermode "Thermal Sensory Analyser TSA-II NeuroSensory Analyzer" and its complement "Vibratory Sensory Analyzer VSA-3000" (Medoc) will be used to assess warm, cold and vibratory detection thresholds, as well as heat and cold painful thresholds. Von Frey monofilaments (Bioseb) will be used to evaluate the mechanical detection threshold. The algometer "Force Ten ™ FDX Digital" (Wagner) will measure the pressure pain threshold. Dynamic mechanical allodynia will be assessed with a standardized brush (SENSELab Brush-05, Somedic). The Neuropen (Owen Mumford) will be used to test the temporal pain summation.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Prud'Homme, MD, PhD, Principal Investigator — Chu de Québec - Université Laval
Locations (2):
- University of Toledo Medical Center, Toledo, Ohio, United States
- CHU de Québec - Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided